CLINICAL TRIAL: NCT01586039
Title: Investigating the Effects of Evening Light Exposure on Melatonin Suppression, Alertness and Nocturnal Sleep.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Biological Illumination, LLC (Industry)
Responsible Party: Principal Investigator, Steven W. Lockley, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 2011-P-002834
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Non-visual Photoreception
Keywords: Melatonin; Sleep; Light; Alertness; Circadian Rhythms

STUDY DESIGN:
Intervention Model Description: Stratified randomized crossover trial. Participants randomized between CFL and LED conditions stratified by light intensity (50 lux and 90 lux).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Compact Fluorescent Light 90 lux (Active Comparator): 90 lux exposure of a commercially available Compact Fluorescent Light (CFL).
  Interventions: Device: Visible light
- Blue-depleted LED light 90 lux (Experimental): 90 lux exposure of a novel LED white light source that is depleted in the short-wavelength visible range (Biological Illumination LCC, FL).
  Interventions: Device: Visible light
- Compact Fluorescent Light 50 lux (Active Comparator): 50 lux exposure of a commercially available Compact Fluorescent Light (CFL).
  Interventions: Device: Visible light
- Blue-depleted LED light 50 lux (Experimental): 50 lux exposure of a novel LED white light source that is depleted in the short-wavelength visible range (Biological Illumination LCC, FL).
  Interventions: Device: Visible light

INTERVENTIONS:
Device: Visible light — We will compare the effects of two light sources, equated for visual stimulus (lux), on multiple non-visual responses to light including melatonin suppression before bedtime. We will compare a 90 lux exposure of a commercially available Compact Fluorescent Light (CFL) with a novel LED white light source that is depleted in the short-wavelength visible range (Biological Illumination LCC, FL).

SUMMARY:
The timing and quality of sleep is governed by environmental and physiologic factors. Environmental factors, especially ambient lighting can impact the circadian system and alter the timing and structure of sleep. Light exposure can also acutely alter neural activation state and impair sleep. These effects all demonstrate marked sensitivity to short-wavelength blue light with maximal sensitivity in the 460-480 nm range. The alerting effects of blue light in the evening persist for at least 3-4 hours after the lights are turned off, and can disturb subsequent sleep. Avoiding these deleterious effects of light exposure prior to sleep on subsequent sleep would be beneficial to sleep quality and potentially health.

The investigators will compare the effects of two light sources, equated for visual stimulus (lux), on multiple non-visual responses to light. The investigators will compare a 90 lux exposure of a commercially available Compact Fluorescent Light (CFL) with a novel LED white light source that is depleted in the short-wavelength visible range (Biological Illumination LCC, FL). In a within-subject design, the investigators will test the hypotheses that exposure to a blue-depleted LED as compared to a CFL exposure at (1) 90 lux or (2) 50 lux will cause significantly:

1. Less melatonin suppression between melatonin onset and bedtime;
2. Less subjective and objective alerting responses before bedtime;
3. Less disruption of nocturnal sleep structure and quality.

ELIGIBILITY:
Inclusion Criteria:

(i) Aged between 18-30 years to reduce the confounding effects of lens aging on the transmission of light to the retina;

(ii) Non-smoking for at least 6 months;

(iii) Healthy (no medical, psychiatric or sleep disorders);

(iv) No clinically significant deviations from normal in medical history, vital signs, physical examination, blood chemistry and hematology, urine chemistry and ECG;

(v) Women of childbearing potential must agree to use an acceptable method of birth control, and must have a negative urine pregnancy test;

(vi) Body mass index of > 18 or < 30 kg/m2;

(vii) No drugs or medication likely to affect sleep or alertness, as determined by the investigators;

(viii) Habitual caffeine consumption < 300mg per day on average;

(ix) Habitual alcohol consumption < 10 alcoholic units per week on average.

Exclusion Criteria:

(i) History of alcohol or substance abuse;

(ii) Positive result on drugs of abuse screening;

(iii) Current or past history of sleep disorders, including but not limited to obstructive sleep apnea, or any significant sleep complaint;

(iv) Psychiatric disorder;

(v) Recent acute or chronic medical disorder, including but not limited to hepatic impairment and severe chronic obstructive pulmonary disease;

(vi) Visual disorder, including but not limited to color blindness, or family history of glaucoma;

(vii) History of intolerance or hypersensitivity to melatonin or melatonin agonists;

(viii) Pregnancy or lactation;

(ix) Shift work;

(x) Transmeridian travel (2 or more time zones) in past 2 months;

(xi) Any other reason as determined by the Principal Investigator.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven W Lockley, Ph.D., Principal Investigator — Brigham and Women's Hospital; Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Compact Fluorescent Light 90 Lux | Blue-depleted LED Light 90 Lux | Compact Fluorescent Light 50 Lux | Blue-depleted LED Light 50 Lux
Started | 8 | 9 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Compact Fluorescent Light 90 Lux | Blue-depleted LED Light 90 Lux | Compact Fluorescent Light 50 Lux | Blue-depleted LED Light 50 Lux | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (1.9) | 24.3 (3.2) | 23.6 (3.1) | 24.8 (3.0) | 24.4 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 16
  Male | 4 | 4 | 4 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 8 | 6 | 7 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 2 | 3 | 6
  White | 8 | 6 | 6 | 4 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Melatonin Suppression
Description: Melatonin suppression is measured as the percentage of melatonin AUC relative to the AUC measured in dim light on the previous day. AUC was calculated during the 6 h of light exposure and the corresponding 6-h interval 24 hours earlier. Higher values indicate more light-induced melatonin suppression.
Time Frame: 6-h constant posture interval of the light exposure
Measure: Mean (Standard Error); unit: Percentage suppression
Arm/Group | Compact Fluorescent Light 90 Lux | Blue-depleted LED Light 90 Lux | Compact Fluorescent Light 50 Lux | Blue-depleted LED Light 50 Lux
Number analyzed (Participants) | 8 | 8 | 8 | 8
Percentage suppression | 71.4 (5.7) | 70.1 (7.2) | 54.3 (5.9) | 32.5 (7.6)
Statistical Analysis 1: Comparison: Compact Fluorescent Light 90 Lux vs Blue-depleted LED Light 90 Lux; Contrasting LED vs. CFL at 90 lux intensity. Melatonin suppression is measured as the percentage of melatonin AUC relative to the AUC measured in dim light on the previous day. Higher values indicate more light-induced melatonin suppression; Test type: Superiority; p = 0.73, t-test, 2 sided — Contrasting LED vs. CFL at 90 lux intensity; Paired t-test
Statistical Analysis 2: Comparison: Compact Fluorescent Light 50 Lux vs Blue-depleted LED Light 50 Lux; Contrasting LED vs. CFL at 50 lux intensity; Test type: Superiority; p = 0.001, t-test, 2 sided — Contrasting LED vs. CFL at 50 lux intensity; Paired t-test

2. Secondary Outcome: Sleep Structure
Description: Sleep efficiency assessed by polysomnography. Sleep efficiency refers to the percentage of time a person sleeps, in relation to the amount of time a person spends in bed trying to sleep. The percentage is calculated by dividing the Total Sleep Time by the Total Time in Bed.
Time Frame: 8-h time in bed immediately following CFL/LED light exposure.
Population: Due to limited financial resources and based on the results of the primary outcome of melatonin suppression in the 90-lux condition, we did not score the PSG data for sleep stage in the 90-lux condition and therefore could not perform an analysis of sleep efficiency. PSG data in one 50-lux condition participant was not collected due to equipment malfunction.
Measure: Mean (Standard Error); unit: % total sleep time of total time in bed
Arm/Group | Compact Fluorescent Light 90 Lux | Blue-depleted LED Light 90 Lux | Compact Fluorescent Light 50 Lux | Blue-depleted LED Light 50 Lux
Number analyzed (Participants) | 0 | 0 | 8 | 7
% total sleep time of total time in bed |  |  | 91.5 (1.0) | 92.4 (1.1)
Statistical Analysis 1: Comparison: Compact Fluorescent Light 50 Lux vs Blue-depleted LED Light 50 Lux; Test type: Superiority; p = 0.19, t-test, 2 sided; Paired t-test

3. Secondary Outcome: Sleep Quality
Description: Self-reported sleep quality was assessed using a post sleep questionnaire. Score on subjective scale range 1-7, higher scores indicate higher sleep quality.
Time Frame: First morning after 8-h time in bed immediately following CFL/LED light exposure.
Population: Post-sleep questionnaires from two participants (each completing once in the "Compact Fluorescent Light 90 lux" condition and once in the "Blue-depleted LED light 90 lux" condition) were not collected due to technical error. As a result n=6 were available for data analysis.
Measure: Mean (Standard Error); unit: Arbitrary units - scale score
Arm/Group | Compact Fluorescent Light 90 Lux | Blue-depleted LED Light 90 Lux | Compact Fluorescent Light 50 Lux | Blue-depleted LED Light 50 Lux
Number analyzed (Participants) | 6 | 6 | 8 | 8
Arbitrary units - scale score | 4.5 (0.2) | 4.6 (0.2) | 4.8 (0.3) | 4.8 (0.2)

4. Secondary Outcome: Subjective Alerting Response
Description: Self-reported sleepiness measured during the light exposure using the Karolinska Sleepiness Scale (KSS). Range of scores 1-9, higher score indicate higher subjective sleepiness. Measures were taken hourly throughout the 6-hour constant posture interval of the light exposure and then averaged to calculate a single value per participant.
Time Frame: 6-h constant posture interval of the light exposure.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Compact Fluorescent Light 90 Lux | Blue-depleted LED Light 90 Lux | Compact Fluorescent Light 50 Lux | Blue-depleted LED Light 50 Lux
Number analyzed (Participants) | 8 | 8 | 8 | 8
Score on a scale | 4.1 (0.2) | 4.3 (0.3) | 4.3 (0.3) | 4.3 (0.3)
Statistical Analysis 1: Comparison: Compact Fluorescent Light 90 Lux vs Blue-depleted LED Light 90 Lux; Test type: Superiority; p = 0.17, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Compact Fluorescent Light 50 Lux vs Blue-depleted LED Light 50 Lux; Test type: Superiority; p = 1.0, t-test, 2 sided; Paired test

5. Secondary Outcome: Objective Alerting Response
Description: Mean reaction time assessed using the 10-minute psychomotor vigilance test. Higher numbers indicate slower reaction times indicating less alertness. Measures were taken hourly throughout the 6-hour constant posture interval of the light exposure and then averaged to calculate a single value per participant.
Time Frame: 6-h constant posture interval of the light exposure
Measure: Mean (Standard Error); unit: Millisecond
Arm/Group | Compact Fluorescent Light 90 Lux | Blue-depleted LED Light 90 Lux | Compact Fluorescent Light 50 Lux | Blue-depleted LED Light 50 Lux
Number analyzed (Participants) | 8 | 8 | 8 | 8
Millisecond | 247.7 (7.2) | 249.7 (7.3) | 229.3 (4.6) | 238.2 (6.7)

ADVERSE EVENTS:
Arm/Group | Compact Fluorescent Light 90 Lux | Blue-depleted LED Light 90 Lux | Compact Fluorescent Light 50 Lux | Blue-depleted LED Light 50 Lux
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/9 | 0/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compact Fluorescent Light 90 Lux (N=8) | Blue-depleted LED Light 90 Lux (N=9) | Compact Fluorescent Light 50 Lux (N=8) | Blue-depleted LED Light 50 Lux (N=8)
Non-serious adverse event (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — gastroenteritis
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Dehydration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No